CLINICAL TRIAL: NCT05741008
Title: Clincal Study of Reduced Target Radiotherapy Based on The Law and Distribution Characteristics of Cervical Lymph Nodes Metastasis in Nasopharyngeal Carcinoma
Brief Title: Clincal Study of Reduced Target Radiotherapy in Nasopharyngeal Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Zhiqiang, Wang, MD,Phd, First Affiliated Hospital of Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021BS005
Record Dates: First submitted 2023-02-11; First posted 2023-02-23 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2023-02

CONDITIONS: Toxicity Due to Radiotherapy; Nasopharyngeal Carcinoma
Keywords: Reduced target; Nasopharyngeal Carcinoma; Radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Reduced target radiotherapy (Experimental): According to our institutional guidelines, GTVnx included the primary tumor volume and the enlarged retropharyngeal nodes, while GTVnd was the volume of involved gross cervical lymph nodes.
  The clinical tumor volume (CTV) includes the primary tumor with potential subclinical disease. The high-risk clinical target volume (CTV1) was defined as the GTVnx plus a 5-mm margin to encompass the high-risk sites of microscopic extension, the whole nasopharynx, retropharyngeal nodal regions and . The low-risk clinical target volume (CTV2) was defined as the whole neck area.(Ib, VIIb, and the commom carotid artery are not included).
  Interventions: Radiation: Target range

INTERVENTIONS:
Radiation: Target range — Compared with conventional radiotherapy, the target dose is unchanged and the CTV2 volume is reduced.

SUMMARY:
To determine whether subtractive radiotherapy can significantly reduce the acute side effects of radiotherapy and improve the quality of life of patients on the basis of ensuring the existing curative effect.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically confirmed nasopharyngeal nonkeratologic carcinoma (differentiated or undifferentiated, i.e., WHO type II or Type III).
2. The clinical stage is TanyN2-3M0, III-IVa (AJCC 8th edition stage).
3. Patients who have not received radiation therapy before.
4. After induction chemotherapy, CR or PR were evaluated by radiography.
5. Age 18-65 years old.
6. ECOG score of 0-1.
7. Good organ function
8. The patient has signed an informed letter and is willing and able to comply with the planned visits, treatment plans, laboratory tests and other research programs.

Exclusion Criteria:

1. Patients with keratinizing squamous cell carcinoma account for only about 5% of the total pathological types, and the sensitivity of radiotherapy is poor compared with the other two types heterogeneous, so nasopharyngeal carcinoma with pathology of keratinizing squamous cells (WHO type I) is excluded.
2. Patients with relapsed and distant metastases.
3. The metastatic lymph nodes are located in the target area (Ib zone, the lateral group of the retropharyngeal lymphatic drainage area (VII), and the cervical lymphatic rainage area The medial border moves from top to bottom from the medial border of the common carotid artery to the lateral border, from the annular cartilage to the superior sternal border, sternoclavicular.The triangular area between the anterior and posterior edges of the medial mastoid muscle and the anterior and lateral border of the jugular arteriovenous sheath and lateral border of the thyroid glanddomain).
4. Nasopharyngeal primary tumor or retropharyngeal metastatic lymph node invasion of oropharynx.
5. Severe heart disease, lung dysfunction, heart function, lung function lower than grade 3 (including grade 3).
6. Those whose laboratory test values do not meet the relevant criteria within 7 days before enrollment.
7. Those who have participated in clinical trials of other drugs within 3 months before treatment.
8. Pregnant or lactating women.
9. Patients assessed by investigators to be unable to cooperate with regular follow-up due to psychological, social, family and geographical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
incidence of acute mucosal ulcers with a toxicity grade 3 or above | up to 6 months
  incidence of acute mucosal ulcers (including those in the oral cavity and pharyngeal wall mucosa) with a toxicity grade 3 or above within 6 months after radiotherapy (that is, between the initiation of radiotherapy to 3 months postradiotherapy) among patients with no recurrence in the reduced-target area

SECONDARY OUTCOMES:
locoregional recurrence-free survival | up to 1 year
  which was defined as the time from enrollment to the occurrence of locoregional recurrence, with the last tumor assessment date serving as the censoring time in the absence of locoregional recurrence
Distant metastasis-free survival | up to 1 years
  The time from date of treatment until date of death due to any cause, assessed up to 1 years.
Overall survival | up to 1 years
  The time from date of treatment until date of death due to any cause, assessed up to 1 years.
Progress Free Survival | up to 1 years
  The time from date of treatment until date of death due to any cause, assessed up to 1 years.
Acute radiation toxicity | up to 3 months
  The injuries after the beginning of radiotherapy include skin, mucosa, pharynx and esophagus, eyes, ears, nervous system, blood system and other organs and tissues，assessed up to 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No